CLINICAL TRIAL: NCT01801683
Title: Application of Evidence Based Medicine in General Practice
Brief Title: Evidence Based Medicine in General Practice
Acronym: EBMINGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split (Other)
Responsible Party: Principal Investigator, Davorka Vrdoljak, PhD, Gp, University of Split
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: Mef01326
Record Dates: First submitted 2013-02-19; First posted 2013-03-01 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Health Knowledge Attitudes and Practice
Keywords: EBM; general practice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: PEARLS (evidence based reports) (Other): Intervention was modified academic detailing method, performed by sixth-year medical students/academic detailers.Each mentor chose two patients from real life who represented diagnostic, therapeutic or prognostic challenge. The students formed an answerable question, using PICO, and wrote report according to PEARLS.
  Interventions: Other: Intervention-using PEARLS
- Control group of GPs (No Intervention): GPs not mentors who do not receive academic detailing intervention using PICO/PEARLS.

INTERVENTIONS:
Other: Intervention-using PEARLS — The intervention applied in this study was the modified academic detailing method, performed by sixth-year medical students as academic detailers. The students qualified for that role because they were taught about EBM in several courses during their undergraduate curriculum. During the family medicine rotation, each GP mentored six students in total. In Split each student visited two mentors for two weeks. In the course of rotation each mentor chose two patients (cases) from real life who represented diagnostic, therapeutic or prognostic challenge. The students' task was to form an answerable question, using the Patient, Intervention, Comparison, Outcome (PICO) scheme, find the best evidence-based answer to that question and to write a brief report according to Practical Evidence about Real Life Situations (PEARLS) pattern. The mentor then reviewed the report and discussed it with the student.
  Other Names: a brief report in accordance with Practical Evidence about Real Life Situations PEARLS
  Arms: Intervention: PEARLS (evidence based reports)

SUMMARY:
Evidence-based medicine (EBM) is the basis of work for physicians- practitioners in all specialties, including family medicine. Various issues in diagnosis, treatment and prognosis appear in daily work with patients and a physician should provide answers based on the best evidence stemming from research. In spite of having access to EBM databases in every GP's office in Croatia, searching and finding answers in consultation with a patient"on the spot" in real time is missing from practice.

OBJECTIVES: To determine GP's knowledge and attitudes about EBM before and after applying modified academic detailing "EBM intervention." provided by sixth- year medical students We assume that GP's knowledge and attitudes about EBM will change as a result of "EBM intervention" applied by students.

DETAILED DESCRIPTION:
STUDY DESIGN:An interventional non-randomized before-and-after study included 98 GPs (49 in the intervention group of mentors and 49 controls) and 174 medical students attending Family Medicine clinical rotations. A telephone survey on knowledge and attitudes towards EBM was conducted among participating physicians before and six months after the rotation. During the rotation, each mentor chose two cases from real life, and the students' task was to form an answerable clinical question, find the evidence-based answer and to write a brief report. The mentor reviewed the report and discussed it with the student.

STUDY SETTING : The sixth year medical students within Family Medicine courses at MedicalSchool in Split, Zagreb and Rijeka have rotations at their mentors' offices. Before arrival of the students, mentors will respond to the questionnaire for physicians prepared for research purposes, and answer the same questionnaire six months after the "EBM intervention." SUBJECTS: mentors /bearers of instructional practices in family medicine constitute the intervention group and the same number of physicians similar in all features to those from the intervention group except that they are not mentors/bearers of instructional practices constitute the control group. The intervention group will be subjected to students' "EBM intervention", and the control will not.

INTERVENTION: The sixth year medical students have practice at their mentors' offices within Family Medicine course. Each mentor chooses two patients / cases from real life, appearing to be diagnostic, therapeutic or prognostic problems in the outpatient work. A student's task is to make a question according to Patient Intervention Comparison Outcome (PICO) scheme, find the best evidence / answer to that question and write a brief report in accordance withPractical Evidence about Real Life Situations PEARL. The report is then brought to the mentor for review and discussion. So, it is a students' "EBM intervention", which will (?) affect the knowledge, attitudes and practice (work style) of a family physician.

MAIN OUTCOME MEASURES: Self-evaluation of knowledge and attitudes after the intervention, which would be a surrogate outcome measure for GP's change in behaviour and work style (adoption of EBM practice).

ELIGIBILITY:
Inclusion Criteria:

All mentors (GPs) mentors of the sixth year medical students

Exclusion Criteria:

Refusal to participate

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
: Self-evaluation of knowledge and attitudes after the intervention, which would be a surrogate outcome measure for GP's change in behaviour and work style (adoption of EBM practice). | February 2013-October 2013 (up to 8 months)

CONTACTS AND LOCATIONS:
Overall Officials: Davorka Vrdoljak, MD Gp PhD, Principal Investigator — University of Split